CLINICAL TRIAL: NCT03983148
Title: Using Motivational Interviewing With Parents in Encouraging Their Children With Cancer to Adopt and Maintain Regular Physical Activity
Brief Title: Motivational Interviewing With Parents to Adopt and Maintain Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HKCH-REC-2019-018
Record Dates: First submitted 2019-06-10; First posted 2019-06-12 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Pediatric Cancer
Keywords: Motivational Interviewing; Parent; Children; Cancer; Physical activity
MeSH Terms: conditions — Neoplasms; Motor Activity | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motivational interviewing (Experimental): Other than usual medical care received by children, their parents in this group will receive three individual, face-to-face interventions on motivational interviewing by a trained registered nurse at baseline, 3-month and 6-month, with each session is about 60 minutes. All sessions of motivational interviewing will be scheduled based on the treatment schedule of the children and conducted in an interview room inside the pediatric oncology unit. A 25-30 minutes semi -structured interview will be conducted for process evaluation at 6-month.
  Interventions: Behavioral: Motivational interviewing
- Placebo control (Placebo Comparator): Other than usual medical care received by children, parents in this group will receive an individual, face-to-face intervention which mimics the time and attention received by those in the experimental group. The intervention includes three sessions of educational talk to parents of children with cancer on healthy diet for cancer patients, adverse effects of cancer treatment, methods to minimize adverse effects.
  Subjects in both groups will receive a booklet developed by the advisory committee, which contains a various kind of physical activities specially designed for children with cancer.
  Interventions: Behavioral: Placebo control

INTERVENTIONS:
Behavioral: Motivational interviewing — There are 3 sessions. Each session is an about 60-minute individual motivational interviewing held by a trained registered nurse. The first session aims to develop an action plan that enables the parents to promote physical activity (PA) for their children. The second session targets to review the adherence to the action plan. The nurse will discuss the progress. In the last session, the aim is to motivate the parents promoting PA for their children in the long run. As such, the benefits of PA throughout the survivorship will be emphasized. And the nurse will work with the parents to identify the resources that can help maintain the designed action plan.
  Arms: Motivational interviewing
Behavioral: Placebo control — Other than usual medical care received by children, parents in this group will receive an individual, face-to-face intervention which mimics the time and attention received by those in the experimental group. The intervention includes three sessions of educational talk to parents of children with cancer on healthy diet for cancer patients, adverse effects of cancer treatment, methods to minimize adverse effects.
  Subjects in both groups will receive a booklet developed by the advisory committee, which contains a various kind of physical activities specially designed for children with cancer.
  Arms: Placebo control

SUMMARY:
Cancer-related fatigue is the most commonly reported symptom among children with cancer and its effect is long-lasting, remaining for years after treatment.Childhood cancer patients undergo chemotherapy and/or radiotherapy that impairs their normal body tissue and fitness. Consequently, cardiorespiratory function and muscle strength decrease, and fatigue is inevitable. More importantly, these complications do not disappear, but continue for months or even years after completion of therapy.

Increasing concern has been placed on the benefits of regular physical activity (PA) among young cancer patients to improve cardiovascular fitness, ameliorate fatigue, and reduce some of the adverse effects of cancer and its treatment. Various studies have shown improvements in quality of life among young patients undergoing cancer treatment by performing regular physical activity. However, the literature review found that most young cancer patients maintain a lower level of PA than before their diagnosis.

A recent study revealed that the current PA levels of Hong Kong young cancer patients were markedly reduced when compared with their pre-morbid situation. Moreover, they were significantly less active in performing physical exercise, and reported lower levels of quality of life than their healthy counterparts. These findings reveal a crucial obligation of health care professionals to advocate the significance of regular PA among young cancer patients.

It is crucial for healthcare to correct misconceptions about PA among parents of children with cancer and advocate the principle of regular PA for their children, with the aim of enhancing their physical and psychological wellbeing and promoting their quality of life. Nevertheless, a large body of evidence has shown that education alone is insufficient or unlikely to change behavior, and healthcare professionals must therefore explore strategies that can actually be effective in helping parents realize the importance of regular physical activities for their children with cancer. Most importantly, healthcare professionals should motivate parents, as the primary caregivers, especially during children's cancer treatment, to take an important role in encouraging their children with cancer to adopt regular PA.

This study aims at testing the effectiveness of using motivational interviewing with parents in encouraging their children with cancer to adopt and maintain regular physical activity.

DETAILED DESCRIPTION:
Despite the mortality rates among cancer patients have been greatly reduced as a result of medical advances in cancer screening and treatment in recent decades, cancer itself and the adverse effects of treatment are still threatening to young cancer patients, with vast destruction in both physical and psychological aspects. In particular, cancer-related fatigue is the most commonly reported symptom among children with cancer and its effect is long-lasting, remaining for years after treatment. Childhood cancer patients undergo chemotherapy and/or radiotherapy that impairs their normal body tissue and fitness. Consequently, cardiorespiratory function and muscle strength decrease, and fatigue is inevitable. More importantly, these complications do not disappear, but continue for months or even years after completion of therapy. All these adverse effects clearly exert both short-term and long-term effects on children and adolescents, severely decreasing their quality of life.

Increasing concern has been placed on the benefits of regular physical activity among young cancer patients to improve cardiovascular fitness, ameliorate fatigue, and reduce some of the adverse effects of cancer and its treatment, including obesity, and osteoporosis. Various studies have shown improvements in quality of life among young patients undergoing cancer treatment by performing regular physical activity. However, the literature review found that most young cancer patients maintain a lower level of physical activity than before their diagnosis.

In a cross-sectional study to examine the physical activity levels and factors that affect their regular physical activity of Hong Kong Chinese childhood cancer survivors, the results revealed a significant decline in physical activity levels in childhood cancer survivors compared with their premorbid situation. In particular, an increasing number of cancer survivors took part in light-intensity activities, whereas a decreasing number of them participated in moderate to vigorous activity.

Another recent study revealed that the current physical activity levels of Hong Kong young cancer patients were markedly reduced when compared with their pre-morbid situation.The amount of time spent in high-intensity activity declined dramatically from 30.3% before diagnosis to only 1.3% during treatment. Moreover, they were significantly less active in performing physical exercise, and reported lower levels of quality of life than their healthy counterparts. These findings reveal a crucial obligation of health care professionals to advocate the significance of regular physical activity among young cancer patients.

There are some reasons to explain why Hong Kong Chinese children undergoing cancer treatment and childhood cancer survivors reported low physical activity levels. Similar to reports in the Western literature, to avoid cancer- or treatment-related fatigue, children are often advised by their parents or even healthcare professionals to take more rest and to reduce their amount of physical activity. In particular, the philosophy of Confucianism focuses on restoring harmony in our bodies to attain health, and this is strongly ingrained in the Hong Kong Chinese population. In this cultural context, cancer and other diseases are regarded as destroying harmony, whereas physical inactivity or rest restore harmony. As a result, childhood cancer patients and survivors are always resting, and they reduce vigorous activities as advised by their parents.

Nevertheless, such recommendation can accelerate fatigue as physical inactivity induces muscle catabolism and atrophy, which in turn may lead to a further decrease in functional capacity. Besides, because of the relatively low body resistance and high susceptibility to infection of children with cancer, many Chinese parents do not allow them near crowded public places, in particular during the seasonal outbreak of influenza, consequently affecting their level of physical activity. Moreover, academic achievement has traditionally been valued above all other forms in Chinese society. This may be due to the attitude commonly held by parents, and most schoolchildren, that academic achievement is related to a better career and brighter future. With this issue in mind, many children with cancer and survivors reported that they were anxious about their academic performance. As a result of suspension from school during the course of treatment and a decreased attention span, coupled with excessive tiredness after remission, they had to make extra efforts to catch up with their studies. Consequently, many did not have time to engage in regular physical activity. In addition, most children with cancer and survivors reported that they lacked encouragement by their parents and role models to follow and learn the physical activities that were appropriate for them to perform. Indeed, parents are influential in affecting the activities that the children performed. In particular, because of sociocultural emphasis on obedience and social conformity, Hong Kong Chinese children are more submissive when compared with Western children. A longitudinal study to examine the relationships between perceived parental psychological control and psychological well-being in Hong Kong Chinese children revealed that parental psychological control may inhibit the development of positive mental well-being and affect emotional life in children.

In sum, the decline in physical activity levels can be attributed to the fact that most Hong Kong Chinese parents overlook the significance of regular physical exercise for their children and misunderstand the effects of physical activity on recovery from cancer and treatment. It is crucial therefore for healthcare to correct misconceptions about physical activity among parents cancer and treatment. It is crucial therefore for healthcare to correct misconceptions about physical activity among parents of children with cancer and advocate the principle of regular physical activity for their children, with the aim of enhancing their physical and psychological well-being and promoting their quality of life. Nevertheless, a large body of evidence has shown that education alone is insufficient or unlikely to change behavior, and healthcare professionals must therefore explore strategies that can actually be effective in helping parents realize the importance of regular physical activities for their children with cancer.

Most importantly, healthcare professionals should motivate parents, as the primary caregivers, especially during children's cancer treatment, to take an important role in encouraging their children with cancer to adopt regular physical activity. There has been an increase in the use of motivational interviewing in lifestyle modifications. In particular, a growing body of evidence support the effectiveness of conducting motivational interviewing with parents to promote different behavioral changes for their children, including weight loss and eating habits. However, there is so far no study to examine whether using motivational interviewing with parents can help promote physical activity among children with cancer.This study aims at testing the effectiveness of using motivational interviewing with parents in encouraging their children with cancer to adopt and maintain regular physical activity.

ELIGIBILITY:
Inclusion Criteria: (Children)

* aged between 9 to 16
* diagnosed with cancer at some time in previous six months and currently admit for cancer treatments
* do not participate in physical exercise and do not intend to start exercising in the next 6 months (pre-contemplation)
* who are able to speak Cantonese and read Chinese.

Exclusion Criteria:(Children)

* children with evidence of recurrence or second malignancies
* those with physical impairment or cognitive and learning problems identified from their medical records

Inclusion Criteria: (Parents)

* must be able to speak Cantonese and read Chinese
* one parent (either father or mother) who should be the main carer for the child with cancer will be selected

Exclusion Criteria: (Parents)

* Parents with emotional or psychiatric disorders, and cognitive and learning problems identified from their medical records

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
Change in levels of physical activity from baseline to 12-month follow-up between intervention and control group | 12-month follow-up
  The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess participants' physical activity levels. It is a one-item scale, scores ranging from 0-2, 3-6 and 7-10 indicate low, moderate and high

SECONDARY OUTCOMES:
Parents' self-efficacy at baseline | baseline
  Self-efficacy of parents will be assessed by asking parents to rate their confidence in engaging their children physically active by using 5-point Likert-type scales ranging from "not confident" to "extremely confident."
Change of parents' self-efficacy from baseline at 6-month follow-up between intervention and control group | 6-month follow up
  Self-efficacy of parents will be assessed by asking parents to rate their confidence in engaging their children physically active by using 5-point Likert-type scales ranging from "not confident" to "extremely confident."
Change of parents' self-efficacy from baseline at 12-month follow-up between intervention and control group | 12-month follow up
  Self-efficacy of parents will be assessed by asking parents to rate their confidence in engaging their children physically active by using 5-point Likert-type scales ranging from "not confident" to "extremely confident."
Children's stages of change at baseline | baseline
  The PASCQ will be used to assess the stages of change about physical activity. This scale contains 4 items and the participants have to answer "yes" or "no" for each of them. With reference to their responses, they are then classified into one of the five stages, including pre-contemplation, contemplation, preparation, action and maintenance.
Change in children's stages of change from baseline at 6-month follow-up between intervention and control group | 6-month follow up
  The PASCQ will be used to assess the stages of change about physical activity. This scale contains 4 items and the participants have to answer "yes" or "no" for each of them. With reference to their responses, they are then classified into one of the five stages, including pre-contemplation, contemplation, preparation, action and maintenance.
Change in children's stages of change from baseline at 12-month follow-up between intervention and control group | 12-month follow up
  The PASCQ will be used to assess the stages of change about physical activity. This scale contains 4 items and the participants have to answer "yes" or "no" for each of them. With reference to their responses, they are then classified into one of the five stages, including pre-contemplation, contemplation, preparation, action and maintenance.
Levels of cancer-related fatigue at baseline | baseline
  The FS-C is designed to assess the severity of fatigue for cancer children aged 9 to 16. This scale contains 14 items which are evaluated on a five-point Likert scale (1= "Not at all"; 2= "A little"; 3= "Some"; 4= "Quite a bit" and 5= "A lot"). The children are asked to indicate their fatigue level over the past 7 days. The possible range of scores is from 14 to 70, with higher scores indicating higher levels of fatigue.
Change in levels of cancer-related fatigue from baseline at 6-month follow-up between intervention and control group | 6-month follow up
  The FS-C is designed to assess the severity of fatigue for cancer children aged 9 to 16. This scale contains 14 items which are evaluated on a five-point Likert scale (1= "Not at all"; 2= "A little"; 3= "Some"; 4= "Quite a bit" and 5= "A lot"). The children are asked to indicate their fatigue level over the past 7 days. The possible range of scores is from 14 to 70, with higher scores indicating higher levels of fatigue.
Change in levels of cancer-related fatigue from baseline at 12-month follow-up between intervention and control group | 12-month follow up
  The FS-C is designed to assess the severity of fatigue for cancer children aged 9 to 16. This scale contains 14 items which are evaluated on a five-point Likert scale (1= "Not at all"; 2= "A little"; 3= "Some"; 4= "Quite a bit" and 5= "A lot"). The children are asked to indicate their fatigue level over the past 7 days. The possible range of scores is from 14 to 70, with higher scores indicating higher levels of fatigue.
Quality of life at baseline | baseline
  The Quality of life of the participants will be measured by the Chinese version of the PedsQL cancer module v. 3.0. All items are evaluated on 5-point Likert scale by which the participants will be asked how much of a problem has been experienced over the last month.
Change in quality of life from baseline at 6-month follow-up between intervention and control group | 6-month follow up
  The Quality of life of the participants will be measured by the Chinese version of the PedsQL cancer module v. 3.0. All items are evaluated on 5-point Likert scale by which the participants will be asked how much of a problem has been experienced over the last month.
Change in quality of life from baseline at 12-month follow-up between intervention and control group | 12-month follow up
  The Quality of life of the participants will be measured by the Chinese version of the PedsQL cancer module v. 3.0. All items are evaluated on 5-point Likert scale by which the participants will be asked how much of a problem has been experienced over the last month.
Levels of physical activity at baseline | baseline
  The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess participants' physical activity levels. It is a one-item scale, scores ranging from 0-2, 3-6 and 7-10 indicate low, moderate and high
Change in levels of physical activity from baseline at 6-month follow-up between intervention and control group | 6-month follow-up
  The Chinese University of Hong Kong: Physical Activity Rating for Children and Youth (CUHK-PARCY) will be used to assess participants' physical activity levels. It is a one-item scale, scores ranging from 0-2, 3-6 and 7-10 indicate low, moderate and high

CONTACTS AND LOCATIONS:
Overall Officials: Ho Cheung William Li, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No